CLINICAL TRIAL: NCT04082507
Title: Alpha-fetoprotein as a Biochemical Marker in Prediction of Placenta Acreta Increta Percreta
Brief Title: Maternal Serum Alpha-fetoprotein Level May Predict the Presence of Morbid Adherent Placenta
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: rasha medhat abdul-hady (Other)
Responsible Party: Sponsor-Investigator, rasha medhat abdul-hady, Lecturer of obstetrics and gynecology, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: AFP_AP
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non_adherent plcenta: placenta separated within 15 minutes after delivery of fetus
- Adherent placenta: placenta dosenot separated within 15 minutes after delivery of fetus
  Interventions: Diagnostic Test: Serum alpha-fetoproteine

INTERVENTIONS:
Diagnostic Test: Serum alpha-fetoproteine — Midtrimesteric serum alpha-fetoprotein mesurment with 2D US and 3D power Doppler with MS US scan .
  Other Names: 2D Ultrasound; 3D power doppler with MS US
  Groups: Adherent placenta

SUMMARY:
The aim of the study is to compare between alpha-fetoproteine as a biological marker and between ultrasound and Doppler in prediction of morbid adherent placenta.

DETAILED DESCRIPTION:
in pregnant women withe previous cesarean section, placenta previa and ultrasonographic finding of an abnormally adherent placenta dose maternal serum alpha-fetoprotein predict prenataly the presence of morbid adherent placenta accurately?

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with history of scarred uterus

  * plcenta previa covering the scar of previous caesarean section as diagnosed by 2DU/S
  * Gestational age from 28wks to full term

Exclusion Criteria:

* pregnant women with fetus with congenital anomalies

  * pregnant women with ovarian swelling
  * pregnant women with medical disease

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 150 pregnant women from 28wk to full term who are attending outpatient clinic and emergency room ain shams university maternal hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Maternal serum alpha-fetoprotein | From 28weeks to 37 weeks
  ng/ml or MOM(Multiple of the median)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt